CLINICAL TRIAL: NCT02817607
Title: Pilot Study to Assess Breast Sensation Before and After Breast Cancer Treatment
Brief Title: Study to Assess Breast Sensation Before and After Breast Cancer Treatment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00068908
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Breast Reconstruction; Ductal Carcinoma In-situ
Keywords: Sensation
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — Biopsy

ARMS (1):
- Surgery (Experimental)
  Interventions: Procedure: Sensory testing and Biopsy

INTERVENTIONS:
Procedure: Sensory testing and Biopsy — Semmes-Weinstein testing: Each breast will be subdivided into 5 regions. This will include the upper 1/3rd, the middle 1/3rd medial and lateral to the nipple areola complex, the lower 1/3rd and the nipple areola-complex. These regions are consistent with the dermatomes described for the breast innervation.
  A cutaneous nerve/skin biopsy is a simple procedure commonly performed on an outpatient setting. The total procedure is expected to take 20 minutes and may be done at the time of surgery as well as 2 and 6 months post operatively either during a revision or at a follow up visit.

SUMMARY:
The purpose of this study is to establish techniques for evaluating breast cutaneous sensation at baseline and following either lumpectomy or mastectomy for breast cancer.

DETAILED DESCRIPTION:
Measuring nerve recovery and breast sensibility has been reported in a limited fashion in the past. A number of studies have assessed patients before and after breast reduction surgery using Semmes-Weinstein monofilaments and found this to be an effective technique. A limited number of studies have been done in patients undergoing mastectomy for breast cancer using these techniques. The main limitation of these existing studies is the lack of prospective measurements before surgery and through time, thus restricting the findings to isolated long-term outcomes. Additionally, no studies have compared patients undergoing mastectomy versus lumpectomy to determine the impact that surgical approach has on breast sensibility.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with ductal carcinoma in-situ (DCIS) or invasive breast cancer
* patients that have been offered lumpectomy or mastectomy for surgical treatment
* patients with a high risk of breast cancer and are pursuing prophylactic mastectomies

Exclusion Criteria:

* metastatic malignancy of any kind
* subjects will not have breast surgery as a portion of their breast cancer care
* between 25 and 65 years old
* subjects with breast implants or a history of prior breast implants
* subjects that have had prior breast reduction surgery
* subjects who have had radiation to one of both breasts in the past
* subjects who cannot give informed consent

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
change in sensory perception score | baseline, time of surgery, 3 months, 6 months
  change in sensory perception will be conducted using paired t-tests or Wilcoxon tests

CONTACTS AND LOCATIONS:
Overall Officials: Scott Hollenbeck, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States